CLINICAL TRIAL: NCT01170260
Title: Alcohol, Marijuana, and Risky Sex: Group Interventions With Detained Adolescents
Acronym: MARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NIAAA RO1 AA013844-05
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Risk Reduction Behavior; Health Behavior; Sexual Behavior; Adolescent Behavior; Cannabis
MeSH Terms: conditions — Risk Reduction Behavior; Health Behavior; Sexual Behavior; Adolescent Behavior; Marijuana Abuse | interventions — Sex; Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Info-only sexual risk reduction (Active Comparator): Corresponding intervention gives information only on STDs/HIV
  Interventions: Behavioral: INFORMATION-ONLY SEXUAL RISK REDUCTION (INFO-ONLY)
- Sex plus alcohol risk reduction (Experimental): Corresponding intervention gives info focusing on sex and alcohol risk reduction only
  Interventions: Behavioral: SEXUAL PLUS ALCOHOL RISK REDUCTION (SRRI+ETOH)
- Sex + alcohol + marijuana risk reduction (Experimental): Corresponding intervention gives info on sex, alcohol, and marijuana risk reduction
  Interventions: Behavioral: SEXUAL + ALCOHOL + MARIJUANA RISK REDUCTION

INTERVENTIONS:
Behavioral: INFORMATION-ONLY SEXUAL RISK REDUCTION (INFO-ONLY) — Intervention includes presentation of STD facts, safe sex activities, condom demonstration, video about sexual decision making, group discussion
  Other Names: INFO-ONLY
  Arms: Info-only sexual risk reduction
Behavioral: SEXUAL PLUS ALCOHOL RISK REDUCTION (SRRI+ETOH) — Intervention includes presentation of STD/alcohol facts, safe sex activities, condom demonstration, video about alcohol/sexual decision making, group discussion
  Other Names: (SRRI+ETOH)
  Arms: Sex plus alcohol risk reduction
Behavioral: SEXUAL + ALCOHOL + MARIJUANA RISK REDUCTION — Intervention includes presentation of STD/alcohol/marijuana facts, safe sex activities, condom demonstration, video about alcohol/marijuana/sexual decision making, group discussion
  Other Names: (SRRI+ETOH+THC)
  Arms: Sex + alcohol + marijuana risk reduction

SUMMARY:
This research is studying behaviors that young people engage in that may place them at risk for contracting a sexually transmitted disease like HIV/AIDS, and what kind of educational program works best to reduce these risky behaviors.

DETAILED DESCRIPTION:
During baseline assessment, a computer questionnaire is administered, including questions about participants' attitudes, beliefs, and behaviors regarding sexual behavior, condom use, and drug use. A saliva sample is provided as well. A "Time-Line Follow-Back" is conducted, noting on which days certain activities occurred, such as sexual intercourse, alcohol use, marijuana use, and cigarette use. A urine sample is also collected in order to test for the STD's chlamydia and gonorrhea (if results are positive, we schedule a meeting with the participant to administer medication to treat the STD).

In the second session, a 3-hour interventional health class is held with groups of same-gender participants. There are 3 different health classes (one focusing just on sex risk reduction, one focusing on sex and alcohol risk reduction, and one focusing on sex, alcohol, and marijuana risk reduction); participants are randomly assigned to one.

Participants are contacted 3 months after the intervention, 6 months after, 9 months after, and 12 months after, in order to meet. These meetings entail completing another Time-Line Follow-Back and completing another questionnaire. At the final 12 month meeting, we collect another urine sample to again test for chlamydia and gonorrhea. As before, if results are positive, we schedule a meeting with the participant to administer medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-18
* Involved in Juvenile Justice System (living in the Detention Center when recruited)

Exclusion Criteria:

* Currently taking anti-psychotics
* Involved in similar intervention-based study (2 similar studies being conducted simultaneously by this lab)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 460 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Juvenile Detention Center (JDC), Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Schmiege SJ, Magnan RE, Yeater EA, Feldstein Ewing SW, Bryan AD. Randomized Trial to Reduce Risky Sexual Behavior Among Justice-Involved Adolescents. Am J Prev Med. 2021 Jan;60(1):47-56. doi: 10.1016/j.amepre.2020.07.009. PMID 33341180
- [Derived] Bryan AD, Magnan RE, Gillman AS, Yeater EA, Feldstein Ewing SW, Kong AS, Schmiege SJ. Effect of Including Alcohol and Cannabis Content in a Sexual Risk-Reduction Intervention on the Incidence of Sexually Transmitted Infections in Adolescents: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2018 Apr 2;172(4):e175621. doi: 10.1001/jamapediatrics.2017.5621. Epub 2018 Apr 2. PMID 29435591

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized to Alcohol Content: Each intervention had identical structure and length (2 hours for intervention, 1 hour for assessments).
- Sex Plus Alcohol Risk Reduction: Corresponding intervention gives info focusing on sex and alcohol risk reduction only
  SEXUAL PLUS ALCOHOL RISK REDUCTION (SRRI+ETOH): Intervention includes presentation of STD/alcohol facts, safe sex activities, condom demonstration, video about alcohol/sexual decision making, group discussio
- Sexual + Alcohol + Cannabis Content: Corresponding intervention gives info on sex, alcohol, and marijuana risk reduction
  SEXUAL + ALCOHOL + MARIJUANA RISK REDUCTION: Intervention includes presentation of STD/alcohol/marijuana facts, safe sex activities, condom demonstration, video about alcohol/marijuana/sexual decision making, group discussion
Period: Overall Study
Arm/Group | Randomized to Alcohol Content | Sex Plus Alcohol Risk Reduction | Sexual + Alcohol + Cannabis Content
Started | 143 | 155 | 162
Completed | 143 | 155 | 162
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Info-only Sexual Risk Reduction | Sex Plus Alcohol Risk Reduction | Sex + Alcohol + Marijuana Risk Reduction | Total
Number analyzed (Participants) | 143 | 155 | 162 | 460
Age, Continuous [Mean (Full Range); unit: years] | 15.85 [15.7 to 16] | 15.82 [15.6 to 16] | 15.78 [15.6 to 16] | 15.81 [15.6 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 78 | 87 | 235
  Male | 73 | 77 | 75 | 225
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 143 | 155 | 162 | 460

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Risky Sexual Behavior Measured for 1 Year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized to Alcohol Content | Sex Plus Alcohol Risk Reduction | Sexual + Alcohol + Cannabis Content
Number analyzed (Participants) | 143 | 155 | 162
Participants | 143 | 155 | 162

ADVERSE EVENTS:
Time Frame: Every 3 months for 1 year
Arm/Group | Randomized to Alcohol Content | Sex Plus Alcohol Risk Reduction | Sexual + Alcohol + Cannabis Content
All-Cause Mortality (participants affected / at risk) | 0/143 | 1/155 | 0/162
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/155 | 0/162
Other Adverse Events (participants affected / at risk) | 0/143 | 0/155 | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes